CLINICAL TRIAL: NCT06642857
Title: Predicting Treatment Response to Immunotherapy Combined with Chemotherapy in Advanced Gastric/gastroesophageal Junction Cancer Based on the Multi-omics Information During Tumor Evolution.
Brief Title: Multi-omics Based Prediction of Treatment Response to Immunotherapy Combined with Chemotherapy in Advanced Gastric/Gastroesophageal Junction Cancer.
Status: Recruiting | Type: Observational
Sponsor: Xiangdong Cheng (Other)
Responsible Party: Sponsor-Investigator, Xiangdong Cheng, Professor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Other Study IDs: IRB-2024-175
Record Dates: First submitted 2024-09-19; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Advanced Gastric Carcinoma; Advanced Gastroesophageal Junction Adenocarcinoma
Keywords: Advanced Gastric Carcinoma; Advanced Gastroesophageal Junction Adenocarcinoma; Chemotherapy combined with immunotherapy; efficacy prediction
MeSH Terms: interventions — Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with advanced gastric cancer: Advanced gastric cancer patients receiving chemotherapy combined with immunotherapy
  Interventions: Other: Peripheral blood, tougue coating, saliva, and feces

INTERVENTIONS:
Other: Peripheral blood, tougue coating, saliva, and feces — Peripheral blood, coating, saliva, and feces on the tongue and clinical data of patients with advanced gastric cancer patients who received chemotherapy combined with immunotherapy will be collected.

SUMMARY:
In this project, based on the information of advanced gastric/gastroesophageal junction cancer in evolution under immunotherapy combined with chemotherapy treatment, we will integrate multi-omics dynamic data to identify essential features that correlate to therapeutic effects of immunotherapy therapy, screen potential molecular markers/dominant microbiota for predicting the efficacy of immunotherapy and establish a multimodal predictive model for patients that benefit from immunotherapy. Our project could provide evidence to predict response to immunotherapy for patients with advanced gastric/gastroesophageal junction cancer and potentially optimize the clinical decision-making about therapy for advanced gastric/gastroesophageal junction cancer.

DETAILED DESCRIPTION:
Main objective: to extract and identify multi omics information tags related to the efficacy of immunotherapy for advanced gastric / gastroesophageal junction cancer

Secondary objective: to construct and validate the efficacy prediction model of chemotherapy combined with immunotherapy for gastric cancer, in order to optimize the scheme decision of advanced gastric cancer treatment

Exploratory purpose: to screen potential molecular markers / dominant flora for predicting the efficacy of immunotherapy in patients with advanced gastric / gastroesophageal junction cancer

ELIGIBILITY:
Inclusion criteria：

* Patients with gastric or gastroesophageal junction adenocarcinoma confirmed by pathology and with advanced or metastatic disease that cannot be resected
* HER2 negative
* Not received any anti-tumor treatment before.
* After evaluation, the treatment plan is chemotherapy combined with immunotherapy.
* Aged 18 to 75 years old, gender is not limited.
* Expected survival time is greater than or equal to 3 months. Exclusion criteria：
* Patients with malignant tumors other than gastric cancer or those with tumors metastasized to the stomach from other sites.
* Patients who have previously received anti-tumor treatments such as surgery, radiotherapy and chemotherapy, targeted therapy or immunotherapy.
* Patients with severe infections.
* Those with a history of mental illness cannot cooperate with the research.
* Patients with severe heart, liver, kidney and other diseases.
* Pregnant or lactating patients.
* HER2 positive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or metastatic gastric or gastroesophageal junction adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective Best Tumor Response | 12 months
  Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Overall Survival | 60 months
  Overall survival is the duration from diagnosis to death. For patients who are alive, overall survival is censored at the last contact.

SECONDARY OUTCOMES:
Progression-free Survival | 36 months
  The period from diagnosis until disease progression or death on study, whichever occurred first.

OTHER OUTCOMES:
Survival rate of 12 month | 12 month from the diagnosis
  The proportion of people who are still alive within 12 month from the diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
We currently have no plans to share individual participant data (IPD) with other researchers.

REFERENCES:
- [Background] Yuan L, Yang L, Zhang S, Xu Z, Qin J, Shi Y, Yu P, Wang Y, Bao Z, Xia Y, Sun J, He W, Chen T, Chen X, Hu C, Zhang Y, Dong C, Zhao P, Wang Y, Jiang N, Lv B, Xue Y, Jiao B, Gao H, Chai K, Li J, Wang H, Wang X, Guan X, Liu X, Zhao G, Zheng Z, Yan J, Yu H, Chen L, Ye Z, You H, Bao Y, Cheng X, Zhao P, Wang L, Zeng W, Tian Y, Chen M, You Y, Yuan G, Ruan H, Gao X, Xu J, Xu H, Du L, Zhang S, Fu H, Cheng X. Development of a tongue image-based machine learning tool for the diagnosis of gastric cancer: a prospective multicentre clinical cohort study. EClinicalMedicine. 2023 Feb 6;57:101834. doi: 10.1016/j.eclinm.2023.101834. eCollection 2023 Mar. PMID 36825238
- [Background] Li MY, Zhu DJ, Xu W, Lin YJ, Yung KL, Ip AWH. Application of U-Net with Global Convolution Network Module in Computer-Aided Tongue Diagnosis. J Healthc Eng. 2021 Nov 18;2021:5853128. doi: 10.1155/2021/5853128. eCollection 2021. PMID 34840700
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525